CLINICAL TRIAL: NCT05340595
Title: Effect of Self-Etch Primer Application on the Bond Failure Rate of a Mandibular Bonded Lingual Retainer
Brief Title: Effect of Primer Application on the Lingual Retainer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Collaborators: Sabahat Yazıcıoğlu (Unknown)
Responsible Party: Principal Investigator, Dr. Fethiye ÇAKMAK ÖZLÜ, Associate Professor, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013/17
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Dental Bonding; Orthodontic Retainers

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): The primer (Transbond XT Primer; 3M Unitek, California) was applied in a thin and uniform coat. Then the adhesive resin (Transbond LR Light Cure Adhesive Paste; 3M Unitek, California) was administered to the lingual surface of the anterior teeth and the lingual retainer was placed in position. The adhesive resin was polymerized from two directions for a total of 20 s using a visible-light curing unit (Hilux 200, Benlioglu Dental Inc., Ankara, Turkey) with an output power of 600 mW/cm2.
  Interventions: Other: Orthodontic retainer bonding
- Study group (Active Comparator): In the study group, the SEP (3M Unitek, Monrovia, California) was used according to the manufacturer's instructions, namely it was administered to the lingual surfaces of the teeth and rubbed for 3 s. Then a gentle burst of dry air was delivered to thin the primer. In the control group, the lingual surfaces of the teeth were etched using 37% phosphoric etchant liquid gel (3M Espe, St Paul, Minnesota, USA) for 30 s, followed by rinsing and drying.
  Interventions: Other: Orthodontic retainer bonding

INTERVENTIONS:
Other: Orthodontic retainer bonding — Self-etch primer (Transbond XT Primer; 3M Unitek, California) was administered to the teeth's lingual surfaces.

SUMMARY:
Background: The aim of this study was to examine the effect of self-etch primer (SEP) application on the bond failure rate of a mandibular bonded lingual retainer over 24 months.

Materials and Methods: After the removal of the orthodontic appliances, the lingual retainers, which were made of six-stranded stainless steel wire 0.0215 inches in diameter, wiil bent and bond onto the lingual surface of all mandibular anterior teeth. The study will performed using a split-mouth design. In the study group, the SEP will be administired to the teeth's lingual surfaces. In the control group, they will etch using 37% phosphoric etchant liquid gel. After etching, the primer wiil be applied. The adhesive resin was applied and the lingual retainer was fitted. The patients will be re-valuated over 24 months. The first bond failures and the amount of adhesive remaining on the tooth will be recorded as the adhesive remnant index (ARI) scores.

The chi-square test will be used to compare the bond failure rates and ARI scores between the groups. The survival rates of the retainers will be estimated using the Kaplan-Meier test. The significance level will P < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who will continue to the retention phase after fixed orthodontic treatment,
2. Presence of all mandibular incisor and canine teeth,
3. Good oral hygiene,
4. No caries,
5. No fractures,
6. Healthy periodontal condition,
7. No restorations,
8. No previous bonded retainer,
9. No traumatic parafunctional habits such as bruxism.

Exclusion Criteria:

-

Ages: 11 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 26 (Actual)
Dates: Start 2014-03-02 (Actual); Primary Completion 2015-11-02 (Actual); Study Completion 2016-07-23 (Actual)

PRIMARY OUTCOMES:
Bond Failure Rate of a Mandibular Bonded Lingual Retainer | 24 months
  Bond Failure Rate of a Mandibular Bonded Lingual Retainer

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Elekdag-Turk S, Isci D, Turk T, Cakmak F. Six-month bracket failure rate evaluation of a self-etching primer. Eur J Orthod. 2008 Apr;30(2):211-6. doi: 10.1093/ejo/cjm119. Epub 2008 Jan 23. PMID 18216373
- [Background] Sfondrini MF, Cacciafesta V, Scribante A, De Angelis M, Klersy C. Effect of blood contamination on shear bond strength of brackets bonded with conventional and self-etching primers. Am J Orthod Dentofacial Orthop. 2004 Mar;125(3):357-60. doi: 10.1016/j.ajodo.2003.09.022. PMID 15014415